CLINICAL TRIAL: NCT03788681
Title: Luteal Phase Support With Estradiol In Poor Responders Undergoing In Vitro Fertilization
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ain Shams Univ
Record Dates: First submitted 2018-12-26; First posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: ICSI
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral estradiol " estradiol valerate (Active Comparator): this group will include ( 85 ) poor responder women undergoing a trial of IVF/ICSI .This group will receive oral estradiol " estradiol valerate " (Cyclo-Progynova® , 2mg , Bayer Schering Pharma Ag , Germany ) from within 24 hours ovum pickup of the cycle.
  Interventions: Drug: Estradiol Valerate
- placebo (Placebo Comparator): this group will include ( 85 ) poor responder women undergoing a trial of IVF/ICSI . This group will receive oral placebo (tablets) from within 24 hours ovum pickup of the cycle
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Estradiol Valerate — oral estradiol " estradiol valerate " (Cyclo-Progynova)
  Arms: oral estradiol " estradiol valerate
Drug: Placebo Oral Tablet — placebo
  Arms: placebo

SUMMARY:
The role of progesterone (P) supplementation in the luteal phase of in vitro fertilization (IVF) cycles is well established world-wide , but the influence of the luteal phase estradiol level on implantation is not clearly defined . There is a significant difference in estradiol levels between fertile and infertile cycles of fertile women who underwent donor insemination.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in this study will have the following criteria : ( 2 of 3 criteria )

  1. advanced maternal age or any other risk factor for POR :

     1. Age ≥35 years
     2. other risk factor of poor responder : ovarian surgery especially in case of endometrioma , chemotherapy, radiotherapy, autoimmune disorders, single ovary, chronic smoking, and unexplained Infertility.
  2. previous poor ovarian response : Number of oocytes at the pickup time 3 or less .
  3. Abnormal ovarian reserve tests :

     1. FSH ≥12 mIu/ml in the early follicular phase .
     2. Estradiol level more than 70 pg/dl in the early follicular phase
     3. Anti-Mullerian hormone (AMH) below 0.5-1.1 ng/ml.
     4. Antral follicle count (AFC) < 5-7 follicles .

Exclusion Criteria:

1. Age >35 with good ovarian response .
2. any intra-uterine pathology can affect receptivity , ( for example ; Sub-mucosal fibroid , intra-uterine adhesions ).
3. Severe male factor infertility.
4. Extended endometriosis (stage 3 or more) .
5. All contraindications for estradiol : venous thrombo-embolism , stroke and breast cancer

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
live birth rate | at least 28 weeks after ET
  the number of deliveries that resulted in a live born neonate

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt